CLINICAL TRIAL: NCT05000814
Title: Study of Cost-effectiveness of the Airway Management and Pulmonary Isolation in Thoracic Surgery Using Standard Double Lumen Tubes vs VivaSight-DL
Brief Title: Study of Cost-effectiveness of the Airway Management in Thoracic Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital General Valencia (Other)
Responsible Party: Principal Investigator, Ruth Martinez Plumed, Principal Investigator, Hospital General Valencia
Other Study IDs: 2021
Record Dates: First submitted 2021-04-13; First posted 2021-08-11 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Brief Description of Focus of Study Instead

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- cDLT: patients using conventional double lumen tube for thoracic surgery
  Interventions: Device: DLT
- VDLT: patients using Vivasight DLT for thoracic surgery
  Interventions: Device: DLT

INTERVENTIONS:
Device: DLT — VDLT versus the use of DLT with fiberoptic bronchoscope

SUMMARY:
The investigators want to carry out a study to determine the role of Doble Lumen Tubes with built-in camera Viva Sight-DL (VDLT) in thoracic surgery. With this study the investigators want to study and enlarge the information in the different surgical approaches, including robotic surgery.

The objective of this study is report a single-center experience using individual data costs to compare the cost effectiveness of VDLT Viva Sight versus the use of conventional Doble Lumen Tubes (cDLT) together with fiberoptic bronchoscope in patients undergoing thoracic surgery, in order to generate information for future decision making related to both devices.

DETAILED DESCRIPTION:
The investigators want to carry out a comparative clinical study on the use of conventional double-lumen endobronchial tubes (cDLT) or video double-lumen endobronquial tubes Vivasight DL (VDLT) during intubation in thoracic lung resection surgery, to study their possible advantages and disadvantages.

This will be a prospective, single-center cohort study of Thoracic Surgery in which the VivaSight-DL (n = 55 patients) or conventional DLT (n = 55 patients) is used for lung isolation in elderly patients (≥ 18 years), thoracic surgery procedures of the "lung resection" type: wedge resection, transegmental resection, lobectomy, bilobectomy or pneumectomy by the different surgical approaches: VATS, robotic surgery and thoracotomy.

The objective of this study is to find out if the use of VDLT reduces the need for fiberoptic bronchoscope (FBS) to verify the positioning of the endobronchial tube during intubation and intraoperatively. Reducing the need for FBS could improve the quality of care provided to the patient and reduce costs to the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patients of legal age (≥18 years).
* Patients who require one-lung collapse in Thoracic Surgery procedures.

Exclusion Criteria:

* Patients with predicted difficult airway.
* Left main bronchus anomalies.
* Previous thoracic surgery.
* BMI> 40.
* Patients with tracheostomy.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing lung resection by thoracotomy, VATS or robotic thoracic surgery.
Sampling Method: Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2023-11-30 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
VDLT reduces the use of fiberoptic bronchoscope | 4 years
  Determine if the use of VivaSight-DL® for lung isolation during lung resections is associated with less need for the use of fiberoptic bronchoscope to check the patient's airway during Thoracic Surgery compared to a conventional double-lumen tube.The cases where VDLT is used and the fiberoptic bronchoscope is necessary will be quantified.
Costs associated with the use of VDLT | 4 years
  * Cost of airway material: includes the use of cDLT as well as the use or not of fiberoptic bronchoscope. The costs of maintenance and cleaning of the same will be included.
  * Cost of the surgical intervention taking the cost / minute of thoracic surgery. Surgeon and surgical assistant, an anesthesiologist, three nurses, a clinic assistant and a caretaker work in these operating rooms. These last two professionals are shared with other operating rooms in the surgical area.
  * Cost of stays in hospitalization room / ICU.
Costs associated with the use of cDLT and fiberoptic bronchoscope | 4 years
  * Cost of airway material: includes the use of cDLT as well as the use or not of fiberoptic bronchoscope. The costs of maintenance and cleaning of the same will be included.
  * Cost of the surgical intervention taking the cost / minute of thoracic surgery. Surgeon and surgical assistant, an anesthesiologist, three nurses, a clinic assistant and a caretaker work in these operating rooms. These last two professionals are shared with other operating rooms in the surgical area.
  * Cost of stays in hospitalization room / ICU.

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Martinez Plumed, Principal Investigator; Manuel Granell Gil, Principal Investigator — Professor, Spanish Society of Anesthesia and Critical Care
Locations (1):
- Ruth Martinez Plumed, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make IPD available.